CLINICAL TRIAL: NCT03733873
Title: Study on the Therapeutic Schedule and Mechanism of Suoquan Mixture Combined With Desmopressin to Children's Monosymptomatic Enuresis
Brief Title: Study on Chinese and Western Medicine in MNE Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Hong Xu，MD.PhD, chief physician, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Suoquan in MNE
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Monosymptomatic Nocturnal Enuresis
Keywords: nocturnal enuresischildren; Chinsese medicine; children; relapse rate
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: group1 desmopressin group2 desmopressin plus Suoquan mixture
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- desmopressin plus Suoquan (Experimental): Drug1. name:desmopressin form:tablet dosage:2-4mg frequency:qn duration:3 months Drug2 name:Suoquan mixture form:liquid dosage:10ml/time frequence:bid duration:3 months
  Interventions: Drug: Desmopressin; Drug: Suoquan
- desmopressin (Active Comparator): name:desmopressin form:tablet dosage:2-4mg frequency:qn duration:3 months
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — take desmopressin for 3 months
  Other Names: Minirin
Drug: Suoquan — take Suoquan mixture for 3 months
  Other Names: Suoquan mixture
  Arms: desmopressin plus Suoquan

SUMMARY:
Monosymptomatic nocturnal enuresis (MNE) is a common pediatric developmental disorder. MNE refers to urinary incontinence in the sleep state in children aged ≥5 years, without other LUT symptoms, and without bladder dysfunction. Its pathogenesis mainly include overnight polyuria, overactive bladder, sleep-arousal dysfunction, genetics, and abnormal secretion of anti-diuretic hormone (ADH). Desmopressin is a synthetic analog of ADH arginine-vasopressin (AVP), which is used to treat central diabetes insipidus and primary nocturnal enuresis (PNE). Desmopressin decreases urine production at night when taken at bedtime. Insufﬁcient ADH secretion at night will contribute to nocturnal polyuria, which is an important cause of NE. Therefore, desmopressin, a synthetic analog of ADH, is frequently used for NE and is an evidence-based therapy (grade ⅠA evidence). Some children, however, have desmopressin resistance and do not achieve the desired treatment goals. What's more,there's a high relapse rate of desmopressin after withdrawing. Suoquan mixture is a Chinese medicine commonly used to treat NE in children. It is composed of Cuscuta, Codonopsis, Psoralea corylifolia Linn ,Astragalus,mantis egg-case and ephedra. It has not only a certain cure rate but also has a lower relapse rate . However there's few evidence could prove that. In this study,the investigators compared the 3 month treatment response and relapse rate (RR) in the following 6 months of desmopressin and desmopressin plus suoquan, and observe if there will be a lower relapse rare in desmopressin plus Suoquan. Moreover, the investigators will try to explore the mechanism of Suoquan mixture in MNE.

ELIGIBILITY:
Inclusion Criteria:

* bedwetting occured ≥2nights/week,last for at least 3 months
* without other LUT symptoms
* without bladder dysfunction.
* no treatment in last 3 months
* signed the consent

Exclusion Criteria:

* had other LUT symptoms
* with bladder dysfunction
* had treatment in last 3 months
* without the consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
the relapse rate of MNE | in 6 months after stopping drugs
  If Suoquan mixture plus desmopressin could reduce the relapse rate of MNE

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, MD.PhD., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No